CLINICAL TRIAL: NCT07316985
Title: Time-Dynamic Study of Gait Variability in Children With Spastic Cerebral Palsy
Brief Title: Time-Dynamic Analysis of Gait Variability in Children With Spastic Cerebral Palsy ( SCP-TIME )
Status: Completed | Type: Observational
Sponsor: LiNa Zhang (Other)
Responsible Party: Sponsor-Investigator, LiNa Zhang, Principal Investigator, Yantai Affiliated Hospital of Binzhou Medical University
Organization: Yantai Affiliated Hospital of Binzhou Medical University (Other)
Other Study IDs: BZMC-SCP-GAIT-2025
Record Dates: First submitted 2025-11-17; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Spastic Cerebral Palsy
Keywords: Gait Variability; Time-Dynamic Analysis; Surface Electromyography; Rehabilitation Training; Motor Function; Children; Spatiotemporal Gait Parameters
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spastic Cerebral Palsy Group: Children diagnosed with spastic cerebral palsy (SCP) according to the Chinese Guidelines for Cerebral Palsy Rehabilitation (2022). Participants aged 3-6 years with Gross Motor Function Classification System (GMFCS) levels I-II performed a 3-minute continuous walking test at a self-selected comfortable speed. Gait and surface electromyography (EMG) parameters were collected to evaluate time-dependent gait variability and muscle activation patterns.
  Interventions: Other: 3-Minute Walking Gait and Surface Electromyography Assessment
- Healthy Control Group: Age-, sex-, and BMI-matched typically developing children without neurological or musculoskeletal disorders. Participants performed the same 3-minute walking test protocol as the SCP group. Gait and surface electromyography data were used as reference values for comparison of spatiotemporal gait parameters and muscle activity changes over time.
  Interventions: Other: 3-Minute Walking Gait and Surface Electromyography Assessment

INTERVENTIONS:
Other: 3-Minute Walking Gait and Surface Electromyography Assessment — Participants performed a 3-minute continuous walking test at a self-selected comfortable speed on a flat surface. Gait parameters were recorded using a portable gait analysis system (IDEEA 3.01, Minisun, USA), and bilateral tibialis anterior and gastrocnemius muscle activity was measured using a Delsys wireless surface EMG system. This standardized assessment procedure was applied to all participants to evaluate time-dependent gait variability and muscle activation patterns.

SUMMARY:
This observational study is designed to investigate the time-dynamic characteristics of gait variability in children with spastic cerebral palsy (SCP). A total of 36 children with SCP and 36 age-, sex-, and BMI-matched typically developing children are recruited from the Children's Rehabilitation Center of the Affiliated Hospital of Binzhou Medical University. Using a portable gait analysis system (IDEEA, Minisun, USA) and a wireless surface electromyography system (Delsys, USA), participants perform a 3-minute continuous walking test at a self-selected comfortable speed. Key spatiotemporal gait parameters and electromyographic root mean square (RMS) values of the tibialis anterior and gastrocnemius muscles are assessed at predefined time points (10 seconds, 1 minute, 2 minutes, and 3 minutes). This study aims to examine temporal changes in gait variability and muscle activation during continuous walking in children with SCP, with the objective of identifying potential time points that may inform the optimization of walking-rest intervals in rehabilitation training.

DETAILED DESCRIPTION:
Spastic cerebral palsy (SCP) is the most common type of cerebral palsy and is characterized by increased muscle tone and impaired motor coordination. Gait variability reflects the dynamic stability and adaptive responses of the locomotor system during walking and is considered an important indicator for functional performance and rehabilitation planning. Understanding how gait parameters and muscle activation patterns evolve over time during continuous walking is essential for designing safe and effective rehabilitation programs for children with SCP. However, the temporal evolution of gait variability during sustained walking in this population remains insufficiently characterized.

This prospective observational case-control study enrolls a total of 72 participants, including 36 children diagnosed with SCP (Gross Motor Function Classification System levels I-II) and 36 typically developing children matched by age, sex, and body mass index. All participants perform a 3-minute continuous walking test at a self-selected comfortable speed on a flat surface.

Spatiotemporal gait parameters are recorded using a portable gait analysis system (IDEEA 3.01, Minisun, USA), while bilateral muscle activity of the tibialis anterior and gastrocnemius muscles is recorded using a Delsys wireless surface electromyography (EMG) system. Gait parameters include step time, cadence, stride length, stance phase, swing phase, gait cycle, and foot lift angle. Surface EMG signals are processed to obtain root mean square (RMS) values as indicators of muscle activation amplitude. Energy expenditure during walking is also estimated using the gait analysis system.

All gait, EMG, and energy expenditure measurements are obtained at predefined time points during the walking task, specifically at 10 seconds, 1 minute, 2 minutes, and 3 minutes after walking initiation. Data analysis is performed using SPSS version 26.0. Between-group comparisons and within-group time-series comparisons are conducted according to data distribution characteristics.

By systematically assessing spatiotemporal gait parameters, muscle activation patterns, and energy expenditure across multiple time points during continuous walking, this study aims to explore the temporal evolution of gait variability in children with spastic cerebral palsy. The results of this study are intended to provide objective data that may inform the development of appropriate walking-rest strategies and individualized rehabilitation programs to support walking safety and functional endurance in children with SCP.

ELIGIBILITY:
Inclusion Criteria:

1. Children diagnosed with spastic cerebral palsy (SCP) according to the Chinese Guidelines for Cerebral Palsy Rehabilitation (2022).
2. Gross Motor Function Classification System (GMFCS) levels I-II.
3. Aged between 3 and 6 years.
4. Able to understand and follow verbal instructions.
5. Informed consent obtained from parents or legal guardians.

Exclusion Criteria:

1. Inability to cooperate with gait or EMG testing.
2. Presence of visual or hearing impairments.
3. History of severe epilepsy or other systemic diseases.
4. Received botulinum toxin or antispastic medication within the past 6 months.
5. Incomplete gait data or failure to complete the walking test.
6. For healthy controls: any neurological, orthopedic, or musculoskeletal disorder, or recent trauma affecting gait.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 3 to 6 years diagnosed with spastic cerebral palsy (SCP) who were receiving rehabilitation therapy at the Children's Rehabilitation Center of the Affiliated Hospital of Binzhou Medical University, and age-, sex-, and BMI-matched healthy children without neurological or musculoskeletal disorders who served as controls.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Step Time | 10 seconds, 1 minute, 2 minutes, 3 minutes
  Step time was captured using the IDEEA 3.01 portable gait analysis system during a 3-minute continuous walking test. Step time values at 10 seconds, 1 minute, 2 minutes, and 3 minutes were compared to quantify temporal changes in gait variability in children with spastic cerebral palsy.

SECONDARY OUTCOMES:
Change in EMG RMS of Tibialis Anterior (µV) | 10 seconds, 1 minute, 2 minutes, and 3 minutes after walking initiation
  Surface EMG signals of the tibialis anterior were collected using a Delsys wireless EMG system during the walking test. RMS amplitude was calculated at 10 seconds, 1 minute, 2 minutes, and 3 minutes to evaluate time-dependent changes in muscle activation.
Change in EMG RMS of Gastrocnemius (µV) | 3-minute continuous walking test
  Surface EMG activity of the gastrocnemius muscle was recorded using the Delsys EMG system. RMS values at each of the four time points were compared to assess fatigue-related reductions in muscle activation during continuous walking.
Change in Energy Expenditure (kCal/min) | 10 seconds, 1 minute, 2 minutes, and 3 minutes after walking initiation
  Energy expenditure was estimated by the IDEEA 3.01 gait system throughout the 3-minute walking task. Temporal changes in metabolic cost were used to assess walking efficiency and fatigue accumulation.
Change in Stride Length (cm) | 10 seconds, 1 minute, 2 minutes, 3 minutes
  Stride length was recorded using the IDEEA 3.01 device at 10 seconds, 1 minute, 2 minutes, and 3 minutes. Changes over time reflect alterations in walking stability and fatigue-related gait adaptations.
Change in Cadence | 10 seconds, 1 minute, 2 minutes, 3 minutes
  Cadence was measured at four time points during the walking test. Temporal differences were analyzed to characterize dynamic gait rhythm changes associated with spastic cerebral palsy.
Change in Stance Phase (% gait cycle) | 10 seconds, 1 minute, 2 minutes, 3 minutes
  The percentage of the gait cycle spent in stance phase was calculated from IDEEA 3.01 data at 10 seconds, 1 minute, 2 minutes, and 3 minutes. Increased stance duration indicates impaired dynamic stability and early fatigue.
Change in Swing Phase | 10 seconds, 1 minute, 2 minutes, 3 minutes
  Swing phase duration as a percentage of the gait cycle was measured at four predefined time points. Reduced swing phase was used as an indicator of compensatory gait adjustments during prolonged walking.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Binzhou Medical University, Binzhou, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including gait parameters, electromyography results, and energy expenditure values, will be available upon reasonable request after publication. Requests can be made to the corresponding author at the Affiliated Hospital of Binzhou Medical University. Data will be shared for academic research purposes only, in compliance with institutional and ethical regulations.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified individual participant data (IPD), including gait parameters, electromyography results, and energy expenditure values, together with the study protocol, statistical analysis plan, and analytic code, will be available beginning 6 months after publication of the primary results and will remain accessible for 3 years. Data will be provided to qualified researchers upon reasonable request and institutional approval through a controlled access process managed by the Affiliated Hospital of Binzhou Medical University.
Access Criteria: Qualified researchers affiliated with academic or non-profit institutions may request access to de-identified individual participant data (IPD) and supporting materials, including the study protocol, statistical analysis plan, and analytic code. Data requests must include a brief proposal describing the intended use and will be reviewed by the Institutional Ethics Committee of the Affiliated Hospital of Binzhou Medical University. Upon approval, data will be shared through a secure institutional data-sharing platform. All shared data will be de-identified and used exclusively for academic research in compliance with institutional and ethical regulations.
URL: https://byfy.cn/Kjc/Index